CLINICAL TRIAL: NCT01057836
Title: Effect of Neck Strength Training on Health-related Quality of Life in Females With Chronic Neck Pain: A Randomized Controlled 1-year Follow-up Study
Brief Title: Effect of Neck Strength Training on Health-related Quality of Life in Females With Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jyväskylä Central Hospital (Other)
Responsible Party: Jari Ylinen, Central Finland Health Care District
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Neck HRQoL
Record Dates: First submitted 2010-01-26; First posted 2010-01-27 (Estimated); Last update posted 2010-01-27 (Estimated); Status verified 2010-01

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Neck strength training (Experimental)
  Interventions: Behavioral: Neck endurance training
- Neck endurance training (Experimental)
  Interventions: Behavioral: Neck endurance training
- Stretching (Active Comparator)
  Interventions: Behavioral: Stretching

INTERVENTIONS:
Behavioral: Neck endurance training
  Arms: Neck endurance training; Neck strength training
Behavioral: Stretching
  Arms: Stretching

SUMMARY:
The purpose of this study is to determine whether intensive one-year neck strength training can enhance health related quality of life in females with chronic neck pain.

ELIGIBILITY:
Inclusion Criteria:

* female
* aged 25 to 53 years
* office worker
* permanently employed
* motivated to continue working
* motivated for rehabilitation
* constant or frequently occurring neck pain for more than 6 months

Exclusion Criteria:

* severe disorders of the cervical spine
* disk prolapse
* spinal stenosis
* postoperative conditions in the neck and shoulder areas
* history of severe trauma
* instability
* spasmodic torticollis
* frequent migraine
* peripheral nerve entrapment
* fibromyalgia
* shoulder diseases (tendonitis, bursitis, capsulitis)
* inflammatory rheumatic diseases
* severe psychiatric illness and other diseases that prevent physical loading
* pregnancy

Ages: 25 Years to 53 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Actual)

PRIMARY OUTCOMES:
15 Dimensional instrument

CONTACTS AND LOCATIONS:
Overall Officials: Jari Ylinen, PhD, MD, Principal Investigator — Central Finland Health Care District
Locations (1):
- Punkaharju Rehabilitation Centre, Punkaharju, Finland

REFERENCES:
- [Derived] Salo PK, Hakkinen AH, Kautiainen H, Ylinen JJ. Effect of neck strength training on health-related quality of life in females with chronic neck pain: a randomized controlled 1-year follow-up study. Health Qual Life Outcomes. 2010 May 14;8:48. doi: 10.1186/1477-7525-8-48. PMID 20465854